CLINICAL TRIAL: NCT01216592
Title: Correlations Between Airway Inflammation, Symptoms and Lung Functions in Patients With Stable Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Airway Inflammation, Symptoms and Lung Function in COPD
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Alberto Papi, Professor, Università degli Studi di Ferrara
Other Study IDs: ISLCOPD01
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Airway inflammation; Symptoms; Lung function; Correlation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum cells.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD
  Interventions: Other: COPD treatment

INTERVENTIONS:
Other: COPD treatment — Patients, will be asked to continue their previous medication (GOLD guidelines) during the study. No interventional change in COPD treatment will be performed during the study.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic inflammatory disease with high prevalence worldwide and with relevant impact on patient-related quality of life, morbidity and mortality. There is evidence that airway inflammation correlates with the severity of the disease and that airway inflammation is further enhanced during exacerbation. However, it is unknown whether daily fluctuation of symptoms or changes in lung function is paralleled by changes in airway inflammation.

DETAILED DESCRIPTION:
Patients will undergo a visit every 7 days during one month (5 visits in total). At each visit airway inflammation (exhaled NO, sputum inflammatory cell count) and lung function will be performed. At home patients will be asked to fill a daily diary for symptom assessment.

ELIGIBILITY:
Inclusion Criteria:

* Post-bronchodilator FEV1/FVC ratio < 70%
* Post-bronchodilator FEV1 < 80%
* Smokers or ex-smoker with pack/years > 15

Exclusion Criteria:

* Atopy
* Asthma
* Concomitant lung diseases (e.g. lung cancer)
* Acute infections of the respiratory tree in the previous 2 months including COPD exacerbation.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate to severe COPD patients (according to GOLD guidelines) will be enrolled in the study
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Correlation between changes in airway inflammation and symptom score | 1 month,
  Correlation between changes in airway inflammation and symptom score will be evaluated

SECONDARY OUTCOMES:
Correlation between changes in airway inflammation and lung function | 1 month
  Correlation between changes in airway inflammation and lung function will be evaluated
Correlations between airway inflammation and symptom scores | 1 month
  Correlation between markers of airway inflammation and symptom score will be performed
Correlations between airway inflammation and lung function | 1 month
  Correlation between markers of airway inflammation and lung function will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Papi, MD, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- Research Centre on Asthma and COPD - Department of Clinical and Experimental Medicine - Section of Respiratory Disease - University of Ferrara, Ferrara, Italy

REFERENCES:
- [Derived] Contoli M, Baraldo S, Conti V, Gnesini G, Marku B, Casolari P, Scrigner P, Morelli P, Saetta M, Spanevello A, Papi A. Airway inflammatory profile is correlated with symptoms in stable COPD: A longitudinal proof-of-concept cohort study. Respirology. 2020 Jan;25(1):80-88. doi: 10.1111/resp.13607. Epub 2019 Jun 28. PMID 31251440